CLINICAL TRIAL: NCT05550610
Title: Evaluation of Mindfulness and Yoga in Basic Combat Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); U.S. Army Training and Doctrine Command (TRADOC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR #2815
Record Dates: First submitted 2022-08-02; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Depressive Symptoms; Anxiety; Sleep; Emotion Regulation; Pain; Military Operations; Cohesion, Social; Mindfulness; Yoga; Leadership; Health, Subjective; Stress; Mood; Musculoskeletal Injury
Keywords: military; basic combat training; soldier; drill sergeant; Mindfulness-Based Attention Training
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation; Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: group randomized trial
Masking Description: All participants were aware whether they were assigned to receive mindfulness and yoga or training as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness and Yoga (Experimental): Mindfulness-Based Attention Training (MBAT) was delivered in 4, 2-hour sessions over 4 weeks. Yoga was delivered 6 days/week, 30 minutes per day.
  Interventions: Behavioral: Mindfulness Based Attention Training (MBAT) and Yoga
- Training as Usual (No Intervention): Training as usual included standard exercises 30 minutes per day during warm-up (15 min) and cool-down (15 min) as part of Army physical readiness training.

INTERVENTIONS:
Behavioral: Mindfulness Based Attention Training (MBAT) and Yoga — Mindfulness-Based Attention Training (MBAT) was delivered in 4, 2-hour sessions over 4 weeks. Participants also completed 15 minutes of group mindfulness practice 6 days/week and received information on embedded practice during the duty day. Yoga was delivered 6 days/week, 30 minutes per day during warm-up (15 min) and cool-down (15 min) as part of Army physical readiness training.
  Arms: Mindfulness and Yoga

SUMMARY:
The present study is a group randomized trial assessing the impact of mindfulness and yoga training on the health, performance, and well-being of soldiers in Basic Combat Training (BCT). Randomization occurred at the platoon level, and platoons received either a combined mindfulness and yoga regimen or training as usual.

DETAILED DESCRIPTION:
This program evaluation assessed a training initiative developed and implemented by the U.S. Army Training and Doctrine Command. Four surveys were conducted with soldiers in all participating platoons over the course of BCT, and two additional surveys were administered with those soldiers in the mindfulness and yoga intervention condition. A follow-up survey was distributed to all participants 6-12 months after BCT. In addition, two surveys were conducted with BCT cadre and drill sergeants. Army data reflecting performance, attrition, and health were also obtained for analysis.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Army soldiers participating in basic combat training from OCT - DEC 2020 at a U.S. Army installation in the southeastern United States.

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1896 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ) Two-Item Version: Change in Scores Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The PHQ-2 is a validated screening tool for depression. The PHQ-2 included a single item assessing impairment in functioning attributable to reported symptoms.
ICD-10 Musculoskeletal Diagnoses: Occurrence Over Time | 0-10 weeks
  ICD-10 musculoskeletal diagnoses (M group) and associated encounter information drawn from U.S. Army records

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD) Two Item Version: Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The GAD-2 is a validated screening tool for anxiety. The GAD-2 included a single item assessing impairment in functioning attributable to reported symptoms.
Insomnia Severity Index (ISI): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks
  The ISI is a validated screening tool for insomnia and sleep-related problems.
Pittsburgh Sleep Quality Index (PSQI) Sleep Quality Item: Change Over Time | 0, 3-4, 6-7, and 9-10 weeks
  A single item from the PSQI was used to assess overall sleep quality.
Defense and Veterans Pain Rating Scale (DVPRS): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The DVPRS is a measure of self-reported pain designed for use in military and veteran populations. The DVPRS was adapted for the present study to assess pain-related interference with training, sleep, mood, and stress.
Patient Health Questionnaire (PHQ-15): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The PHQ-15 is a validated measure of a range of patient health outcomes. Ten items from the PHQ-15 were used to assess physical pain and assorted medical symptoms.
Mental Toughness Inventory (MTI): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The MTI is a measure of mental toughness and resilience. Eight items from the MTI were used in the present evaluation: Four items assessed mental toughness during stressful events, and four items assessed mental toughness following stressful events.
Multidimensional Assessment of Interoceptive Awareness (MAIA): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The MAIA is a measure of interoceptive awareness and mindfulness-related constructs. Ten items from the MAIA were used in the present evaluation: Six items assessed the capacity to not self-distract, and four items assessed capacity for self-regulation.
Five Facet Mindfulness Questionnaire (FFMQ): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks
  The FFMQ is a measure of engagement in mindful awareness.
Brief Difficulties in Emotion Regulation Scale (DERS): Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  The Brief DERS is a shortened version of a validated measure assessing ability to manage difficult emotions. Subscales assessed difficulties with emotional awareness, impulse control, and engaging in goal-directed behavior.
Attitudes toward Mindfulness Training: Change Over Time | 0, 3-4, 6-7, and 9-10 weeks
  Four items developed for the current evaluation were used to assess perceived acceptability and utility of mindfulness training.
Overall Health: Change Over Time | 0, 3-4, 6-7, and 9-10 weeks; 6-12 month follow-up
  A single item was used to assess self-rated health.
Indiscipline: Occurrence Over Time | 3-4, 6-7, and 9-10 weeks
  Seven items developed for the current evaluation were used to assess behaviors that reflect indiscipline and consequences experienced as a result of indiscipline.
Satisfaction with Yoga or Preparatory and Recovery Drills: Change Over Time | 3-4, 6-7, and 9-10 weeks
  Eleven items developed for this evaluation were used to assess satisfaction with yoga intervention and preparatory and recovery drills.
Unit Cohesion: Change Over Time | 3-4, 6-7, and 9-10 weeks
  A validated three-item measure was used to assess unit cohesion.
Self-Reported Medical Visits: Occurrence Over Time | 0, 3-4, 6-7, and 9-10 weeks
  A single item measure developed for this evaluation was used to assess frequency of medical visits.
Self-Reported Pain: Change Over Time | 0, 3-4, 6-7, and 9-10 weeks
  Three items were developed for this evaluation assessing the frequency of pain, level of pain, and chronicity of pain.
Impact of Injury on Training: Change Over Time | 3-4, 6-7, and 9-10 weeks
  Eight items developed for the present evaluation were used to assess disruption in training due to injury, trainee response to injury, and outcomes associated with experience of injury.
Use of Mindfulness following Training | 6-12 month follow-up
  Twenty-five items were developed for the present evaluation to assess use of mindfulness and attitudes towards mindfulness practice following basic combat training.
Use of Yoga or Preparatory and Recovery Drills (PRT) following Training | 6-12 month follow-up
  Twenty-three items were developed for the present evaluation to assess use of yoga/PRT drills and attitudes towards yoga/PRT drills following basic combat training.
Use of Mindfulness and Yoga Resources following Training | 6-12 month follow-up
  Nine items were developed for this evaluation to assess receipt and use of mindfulness and yoga resources following training.
Use of Mindfulness during Training: Change Over Time | 3-4 weeks; 9-10 weeks
  Thirteen items were developed for this evaluation to assess use of MBAT during basic combat training.
Perceived Drill Sergeant Support for Mindfulness during Training: Change Over Time | 3-4 weeks; 9-10 weeks
  Six items were developed for this evaluation to assess trainees' perception of drill sergeant support for MBAT during basic combat training.
Drill Sergeant Leadership: Change Over Time | 3-4 weeks; 9-10 weeks
  Nine items were used to assess participants' perceptions of the quality of drill sergeant's leadership and instruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Jackson, Fort Jackson, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data are available for research upon reasonable request and completion of institute-related agreements.

REFERENCES:
- [Background] Nassif TH, Start AR, Toblin RL, Adler AB. Self-reported mindfulness and soldier health following a combat deployment. Psychol Trauma. 2019 May;11(4):466-474. doi: 10.1037/tra0000413. Epub 2018 Nov 5. PMID 30394773
- [Background] Janssen M, Heerkens Y, Kuijer W, van der Heijden B, Engels J. Effects of Mindfulness-Based Stress Reduction on employees' mental health: A systematic review. PLoS One. 2018 Jan 24;13(1):e0191332. doi: 10.1371/journal.pone.0191332. eCollection 2018. PMID 29364935
- [Background] Domingues RB. Modern postural yoga as a mental health promoting tool: A systematic review. Complement Ther Clin Pract. 2018 May;31:248-255. doi: 10.1016/j.ctcp.2018.03.002. Epub 2018 Mar 10. PMID 29705463
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] Jha AP, Denkova E, Zanesco AP, Witkin JE, Rooks J, Rogers SL. Does mindfulness training help working memory 'work' better? Curr Opin Psychol. 2019 Aug;28:273-278. doi: 10.1016/j.copsyc.2019.02.012. Epub 2019 Mar 6. PMID 30999122
- [Background] Zanesco AP, Denkova E, Rogers SL, MacNulty WK, Jha AP. Mindfulness training as cognitive training in high-demand cohorts: An initial study in elite military servicemembers. Prog Brain Res. 2019;244:323-354. doi: 10.1016/bs.pbr.2018.10.001. Epub 2018 Nov 27. PMID 30732844
- [Derived] Nassif TH, Gutierrez IA, Smith CD, Jha AP, Adler AB. The Effect of a Combined Mindfulness and Yoga Intervention on Soldier Mental Health in Basic Combat Training: A Cluster Randomized Controlled Trial. Depress Anxiety. 2023 Dec 1;2023:6869543. doi: 10.1155/2023/6869543. eCollection 2023. PMID 40224611
- [Derived] Smith CD, Gutierrez IA, Nassif TH, Jordan KL, Taylor KM, Jha AP, Adler AB. Impact of mindfulness training and yoga on injury and pain-related impairment: a group randomized trial in basic combat training. Front Psychol. 2023 Oct 6;14:1214039. doi: 10.3389/fpsyg.2023.1214039. eCollection 2023. PMID 37868598